CLINICAL TRIAL: NCT03576053
Title: En Mekanistisk undersøgelse af Interaktioner Imellem Det Thermoceptive og Det Pruriceptive Sensoriske System
Brief Title: A Mechanistic Evaluation of the Interactions Between Thermoceptive and Pruriceptive Sensory Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Daniele Riccio, Principal investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: N-20180035
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Itch; Thermal Stimulation; Histamine; Cowhage; Serotonine
MeSH Terms: conditions — Pruritus | interventions — Lidocaine; Histamine; Serotonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only the third sub-study is conducted in a double-blind manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Histamine+cowhage+heat (Experimental)
  Interventions: Other: Histamine; Other: Cowhage; Other: Heat stimulation
- Histamine+cowhage+serotonin+pre-heating (Experimental)
  Interventions: Other: Histamine; Other: Cowhage; Other: Pre-heating; Other: Serotonin
- lidocaine and saline+heat (Placebo Comparator)
  Interventions: Drug: Lidocaine; Other: Heat stimulation

INTERVENTIONS:
Drug: Lidocaine — Lidocaine intradermal injection
  Arms: lidocaine and saline+heat
Other: Histamine — Skin Prick Test with Histamine
  Arms: Histamine+cowhage+heat; Histamine+cowhage+serotonin+pre-heating
Other: Cowhage — Manually skin insertion of cowhage spicules
  Arms: Histamine+cowhage+heat; Histamine+cowhage+serotonin+pre-heating
Other: Heat stimulation — Short heat stimulation
  Arms: Histamine+cowhage+heat; lidocaine and saline+heat
Other: Pre-heating — Mild skin pre-heating
  Arms: Histamine+cowhage+serotonin+pre-heating
Other: Serotonin — Serotonin electrophoresis
  Arms: Histamine+cowhage+serotonin+pre-heating

SUMMARY:
The purpose of this human experimental study is to evaluate the pattern of itch intensity over time in response to strong, short-term heat stimulation in two different models of histamine and cowhage-induced itch. Moreover, the purpose is to evaluate the effect of mild pre-heating of the skin in human experimental models of histamine, cowhage and serotonin. Finally, we want to investigate the effect of short-term intense heat stimulation on previously anesthetized skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-60 years
* Able to speak and understand English

Exclusion Criteria:

* Suffering from chronic disease
* Pregnancy or lactation
* Prior experience of adverse effects from anaesthetic, specifically Lidocaine
* Drug addiction defined as the use of cannabis, opioids or other drugs - 5 -
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* Current use of medications that may affect the trial
* Active skin diseases
* Active participation in other experiments currently ongoing or within the last 14 days
* Tattoos on volar forearms that will interfere with local skin measurements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
eVAS Itch | 10 minutes
  Electronic Visual Analog Scale for itch sensation. 0-100 scale, it measures the self-estimated itch the subject experience on a scale where 0 correspond to "No itch" and 100 "Worst itch imaginable".
Skin temperature | 5 seconds
  Infrared skin thermometer
eVAS Pain | 10 minutes
  Electronic Visual Analog Scale for pain sensation. 0-100 scale, it measures the self-estimated pain the subject experience on a scale where 0 correspond to "No pain" and 100 "Worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Riccio, MSc, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No